CLINICAL TRIAL: NCT05712187
Title: A Randomized, Double-Blind, Placebo-Controlled Study of ALTO-100 With an Open-Label Extension in Adults With Major Depressive Disorder
Brief Title: Phase 2b Study of ALTO-100 in MDD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alto Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTO-100-201
Record Dates: First submitted 2022-12-24; First posted 2023-02-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2024-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALTO-100 (Experimental): Participants will receive ALTO-100 tablet twice daily, from Day 1 to Day 42 in double blind (DB) treatment period. Eligible participants who will enter the open label (OL) treatment period will receive ALTO-100 tablet twice daily from OL baseline until the end of OL period/early termination visit (Up to 7 weeks).
  Interventions: Drug: ALTO-100
- Placebo DB (Placebo Comparator): Participants will receive matching placebo tablet twice daily, from Day 1 to Day 42 in double blind (DB) treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALTO-100 — ALTO-100 tablet BID
  Arms: ALTO-100
Drug: Placebo — Placebo tablet BID
  Arms: Placebo DB

SUMMARY:
The purpose of this study is to determine efficacy differences between ALTO-100 and placebo, used either as monotherapy or adjunctively to an antidepressant, related to patient characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of moderate to severe major depressive disorder (MDD)
* At baseline, either not taking an antidepressant medication, or currently taking a single SSRI, SNRI, mirtazapine, or bupropion for at least 6 weeks with no dose modifications in the past 2 weeks
* Willing to comply with all study assessments and procedures
* Must not be pregnant or breastfeeding at time of enrollment or throughout study

Exclusion Criteria:

* Evidence of unstable medical condition
* Diagnosed bipolar disorder, psychotic disorder, or dementia
* Current moderate or severe substance use disorder
* Has a history of hypersensitivity or allergic reaction to ALTO-100 or any of its components/excipients
* Concurrent or recent participation in another clinical trial for mental illness involving an investigational product or device

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
To assess efficacy of ALTO-100 versus placebo on symptoms of MDD in a pre-defined subgroup of participants as measured by the change from Day 1 to Week 6 on the Montgomery-Åsberg Depression Rating Scale (MADRS) total score. | Change assessed from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
To assess efficacy of ALTO-100 versus placebo for symptoms of MDD in a pre-defined subgroup of participants who are taking ALTO-100 as monotherapy for MDD as measured by the change from Day 1 to Week 6 on the MADRS total score. | Change assessed from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 versus placebo on symptoms of MDD in all randomized participants as measured by the change from Day 1 to Week 6 on the Montgomery-Åsberg Depression Rating Scale (MADRS) | Assessed 4 times over a 6 week interval, from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 versus placebo for MDD as measured by the change from Day 1 to Week 6 in Clinician Global Impression Scale-severity (CGI-S). | Assessed 4 times over a 6 week interval, from Day 1 to Week 6
  The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of illness exhibited by a participant, rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 vs placebo for MDD as measured by the change from Day 1 to Week 6 in response (>50% improvement from baseline) and remission (total MADRS score of <10) rates based on the Montgomery-Åsberg Depression Rating Scale (MADRS) | Assessed 4 times over a 6- week interval, from Day 1 to Week 6
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
To assess efficacy of ALTO-100 versus placebo for MDD as measured by the change from Day 1 to Week 6 in Patient Health Questionnaire, 9 item (PHQ-9). | Assessed 4 times over a 6- week interval, from Day 1 to Week 6
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders-5th edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4- point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
To evaluate the safety of ALTO-100 during both the OL and DB periods of the study as measured by the assessment of the incidence, severity, and relatedness of Adverse Events. | Assessed from Day 1 to Week 13
  Incidence, severity, and relatedness of Adverse Events.
To evaluate the safety of ALTO-100 during both the OL and DB periods of the study as measured by the assessment of Heart Rate. | Assessed from Day 1 to Week 13
  Assessment of Heart Rate.
To evaluate the safety of ALTO-100 during both the OL and DB periods of the study as measured by the assessment of Blood Pressure. | Assessed from Day 1 to Week 13
  Assessment of Blood Pressure.
To evaluate the safety of ALTO-100 during both the OL and DB periods of the study as measured by the assessment of Weight. | Assessed from Day 1 to Week 13
  Assessment of Weight.
To evaluate the safety of ALTO-100 during both the OL and DB periods of the study as measured by the assessment of suicidality with the Concise Health Risk Tracking Self-Report,12 item scale (CHRT-SR12). | Assessed from Day 1 to Week 13
  The CHRT is a brief, self-report measure that systematically assesses both suicidal thinking and associated thoughts that may indicate the propensity for suicidal acts. The CHRT-SR12 is a 12 item scale. The patient assigns a score of 0-4 for each item of the scale, allowing for a total score of 0 to 48, with the higher score signifying more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Savitz, MD, PhD, Study Director — Alto Neuroscience
Locations (34):
- United States (34):
  - Site 174, Birmingham, Alabama
  - Site 173, Huntsville, Alabama
  - Site 136, Chandler, Arizona
  - Site 139, Little Rock, Arkansas
  - Site 141, Costa Mesa, California
  - Site 118, Fresno, California
  - Site 181, Imperial, California
  - Site 182, Oceanside, California
  - Site 188, Oceanside, California
  - Site 179, Rancho Cucamonga, California
  - Site 116, Sacramento, California
  - Site 185, Centennial, Colorado
  - Site 186, Brooksville, Florida
  - Site 204, Jacksonville, Florida
  - Site 205, Orlando, Florida
  - Site 212, Tampa, Florida
  - Site 213, Tampa, Florida
  - Site 137, Carmel, Indiana
  - Site 151, Baltimore, Maryland
  - Site 108, Jackson, Mississippi
  - Site 171, Jackson, Mississippi
  - Site 142, Lincoln, Nebraska
  - Site 144, Las Vegas, Nevada
  - Site 178, Albuquerque, New Mexico
  - Site 184, Brooklyn, New York
  - Site 180, New York, New York
  - Site 210, New York, New York
  - Site 175, Westlake, Ohio
  - Site 157, North Charleston, South Carolina
  - Site 183, Memphis, Tennessee
  - Site 147, Fort Worth, Texas
  - Site 120, Houston, Texas
  - Site 172, Houston, Texas
  - Site 121, Draper, Utah

IPD SHARING:
Plan to Share IPD: No